CLINICAL TRIAL: NCT04454502
Title: Analysis of the Effects of Oral Colostrum Administration in Very Low Birth Weight Premature Infants Who Cannot be Fed Orally on the Breastfeeding
Brief Title: Analysis of the Effects of Oral Colostrum Administration in Premature Infants on the Breastfeeding
Acronym: Oral colostrum
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, Özge Karakaya Suzan, research asistant, Sakarya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: oral colostrum
Record Dates: First submitted 2020-06-22; First posted 2020-07-01 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Oral Colostrum Administration in Very Low Birth Weight Premature Infants
Keywords: very low birth weight premature infants,; oral colostrum administration,; breastfeeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: : Randomized Controlled Trial
Who Masked: Outcomes Assessor
Masking Description: Single-blind (researchers are not blind) randomization will be provided since the mothers will be provided with education on the importance of oral colostrum administration and milking techniques by the researchers. The statistician was also blinded for the data analysis purpose
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): In the first stage of data collection, the information in the "Mother-Preterm Introductory Information Form" study and control groups before colostrum administration, and the information in "Preterm Follow-up Form" including questions related to physiological parameters, body measurements and nutrition will be obtained. In the second stage, oral colostrum, will be administered once every 3 hours and for at least 5 days until the newborn begins oral feeding. In accordance with the oral colostrum protocol, a total of 0.2ml colostrum will be administered in approximately 1 minute for infants weighing between 1001-1500 g. The third stage, the effectiveness of the first breastfeeding will be evaluated by the observers in experimental group using the Bristol Breastfeeding Assessment Tool. In the last stage, one week after the first breastfeeding sucking / breastfeeding experience will be evaluated again.
  Interventions: Other: Oral colostrum administration
- Control Groups (No Intervention): The infants in the control group will be followed up by oral care with sterile physiological saline in routine care of the service

INTERVENTIONS:
Other: Oral colostrum administration — In accordance with the oral colostrum protocol, a total of 0.2ml colostrum will be administered into the cheek and on the tongue for the infants weighing between 1001-1500 g.
  Arms: Experimental

SUMMARY:
In the literature, it is emphasized that oral colostrum administration in very low birth weight infants supported the immune development of the premature newborn, contributed to the development of oral microbiota and reduced the length of hospital stay (Manzoni 2011; Pammi 2011; Zhang 2017; Moreno-Fernandez 2018; Rodriguez 2009). However, there was no source answering the question of how both the mother and the infant are affected by oral colostrum administration in very low birth weight infants. Based on the studies indicating that premature infants distinguished their mother's milk smell and taste (Lecanuet and Schoal, 1996; Aoyama et al. 2010), it was aimed to find answers to the questions of whether this administration in infants without oral intake had positive effect on the success of breastfeeding.

Research Hypotheses:

H0: Oral colostrum administration in very low birth weight premature infants who cannot be fed orally has no effect on breastfeeding.

H1: Oral colostrum administration in very low birth weight premature infants who cannot be fed orally affects the success of breastfeeding

DETAILED DESCRIPTION:
Background: Premature newborns are physiologically and structurally different from mature newborns, and these differences also bring along many health problems. Healthy growth and neurodevelopmental needs of premature infants are evolutionarily met by providing breast milk, which is a unique and natural food with excellent content. The importance of breast milk in the nutritional management of premature and risky newborns has been well documented by the American Academy of Pediatrics (American Academy of Pediatrics. 2012), and colostrum with rich content especially in breast milk is the perfect first immunostimulant in infants. In the literature, it is emphasized that oral minimal colostrum administration in very low birth weight infants supports the development of immunity, contributes to the development of oral microbiota and reduces the length of hospital stay (Manzoni 2011; Pammi 2011; Zhang 2017; Moreno-Fernandez 2018; Rodriguez et al. 2009; Rodriguez et al. 2010).

In the intrauterine period, while the development of the sense of smell is completed at gestational weeks 26-28, the development of the sense of taste is completed at week 18. The fact that premature newborn is physically and neurologically insufficient after birth, and the failure of environmental factors to meet the sensory needs (smell, taste, touch, sight, hearing) in the intensive care environment outside the safe intrauterine environment during the critical period negatively affect the newborn. The sense of smell is related to the sense of taste and is a rapidly developing "chemical" sense. In the literature, it is reported that familiar and pleasant tastes and smells facilitate the psychophysiological adaptation of premature newborns to the first environment and contribute to mother-infant attachment (Lipchock et al. 2011; Henderson 2011). The fats secreted from montgomery bodies (small mounds on the areola) in the newborn's mother's breast have the same chemical structure and smell of the amniotic fluid. This special similarity supports the sensory development of the newborn and also helps the newborn to find and grasp the mother's breast (Henderson 2011; Mennella and Ventura 2011). In the studies, it is reported that the taste and smell of breast milk have effects on increased sucking movements of the newborn, early transition to oral feeding and soothing (Aoyama et al. 2010; Bingham, Abassi and Sivieri 2003). It is considered that there are many factors that affect the breastfeeding experience, and that one of the most important of these experiences is the newborn's gaining sensory experience for the senses of smell and taste until the first breastfeeding experience. Based on the studies indicating that premature infants distinguish their mother's milk smell and taste (Lecanuet and Schoal, 1996; Aoyama et al. 2010), it is considered that the newborns will positively affect the breastfeeding with the oral colostrum administration. The aim of this study was to analyze the effect of oral (oropharyngeal) colostrum administration in very low birth weight premature infants (between 1000-1500 gr) who cannot be fed orally on the success of breastfeeding.

Method: This is a randomized controlled experimental study. All very low birth weight infants born to primiparous mothers hospitalized in the Neonatal Intensive Care Unit of Sakarya University Training and Research Hospital, Ministry of Health between February and November 2020 will constitute the population of the study. The sample of the study was calculated in accordance with the intervention group selection criteria and by performing power analysis. Power analysis was performed using G*Power (v3.1.7) program in order to determine sample size. The effect range value was taken as 0.70 as the method used in cases where it is unknown how many units difference is significant between the groups. In cases where Type 1 error probability (α) was 0.05 (at a confidence level of 95%), at a power level of 80% and the effect range was 0.70, the study was planned with a total of 68 mothers, including 34 mothers women for each group. In the study, randomization will be determined by the urn method. The urn method is used as a method equivalent to full randomization. In this method, two parameters such as α and β are mentioned. These parameters refer to balls in two different colors, red and white. α can be white or red, and β will be the exact opposite of them. One of the balls is randomly selected and if the selected ball is white, the individual is allocated into group α, and if it is red, then the individual is allocated into group β. This process is repeated in each allocation (Kanık et al. 2011). In the study, the red colored ball constituted the study group and the white colored ball constituted the control group. In the case of an infant who meets the sampling criteria, these balls prepared by the researcher will be placed in a black pouch and a nurse currently working in the unit will be asked to make a choice with her eyes closed. The infant will be allocated into the study or control group according to the color of the selected ball. Thus, the infants will be randomly allocated into both groups.. The sample of the study will be randomly allocated into two groups: the intervention group will be administered with oral colostrum, and the other group, which was the control group, will be followed up by oral care with sterile physiological saline in routine care of the service. Single-blind (researchers are not blind) randomization will be provided since the mothers will be provided with education on the importance of oral colostrum administration and milking techniques by the researchers. The statistician was also blinded for the data analysis purpose. Data collection will be conducted in five stages. In the first stage of data collection, the information in the "Mother-Preterm Introductory Information Form" including socio-demographic characteristics in the study and control groups before colostrum administration, and the information in "Preterm Follow-up Form" including questions related to physiological parameters, body measurements and nutrition will be obtained. In the second stage, oral colostrum, which was initiated when the neonatologist determined that the newborn in the study group was stable, will be administered once every 3 hours and for at least 5 days until the newborn begins oral feeding. In accordance with the oral colostrum protocol, a total of 0.2ml colostrum will be administered in approximately 1 minute for infants weighing between 1001-1500 g. The infants in the control group will be followed up in routine service care. In the third stage, the information in the "Preterm Follow-up Form" will be obtained after oral colostrum administration in the study group. The same data will be obtained from the control group simultaneously with the study group. In the fourth stage, the effectiveness of the first breastfeeding will be evaluated by the observers in both groups using the Bristol Breastfeeding Assessment Tool. In the last stage, one week after the first breastfeeding sucking / breastfeeding experience will be evaluated again. In the evaluation of data, statistical analyses will be performed using the SPSS package program. The Kolmogorov-Smirnov (K-S) test will be used for normality. In order to determine whether there is a difference in the dependent variables compared to independent variables, the independent group t-test will be used if the distribution is normal in independent variables with two options, and Mann Whitney-U test will be used if distribution is not normal. The results will be evaluated at a confidence level of 95% and at a level of significance of p<0.05.

ELIGIBILITY:
İnclusive criteria

* Newborn's body weight between 1001-1500gr
* Newborn being premature (>28 and < 32 GW)
* Being admitted to the neonatal intensive care unit within the first 24 hours after birth
* Absence of congenital anomaly (craniofacial abnormality such as cleft palate, cleft lip, paralysis of facial muscles) in the newborn
* Absence of any diagnosed gastrointestinal, neurological and genetic disease (necrotizing enterocolitis, third and fourth level intracranial hemorrhage (ICH), periventricular leukomalacia, hydrocephalus, down syndrome, omphalocele, gastroschisis, short bowel syndrome and other diseases) in the newborn
* Absence of congenital heart disease requiring surgical treatment in the newborn
* Absence of Oral feeding of the newborn (Nasogastric/orogastric or trophic feeding can be done)
* Non-contraindication of the mother's milk to her infant
* Absence of the mother's diagnosed psychiatric story
* Mother's openness to communication and cooperation
* Mother's volunteering to participate in the study
* Bringing sufficient colostrum for administration by the mother
* Mother being literate
* Mother being primiparous and having single infant
* Mother's age above 18 years Exclusive criteria
* Newborn being SGA and LGA
* Mother's not coming to breastfeed her infant between two breastfeeding follow-ups

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 68 (Estimated)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2021-08-01 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in The Bristol Breastfeeding Assessment Tool | The difference between the first Breastfeeding Day and the breastfeeding activity one week after the first breastfeeding
  The Bristol Breastfeeding Assessment Tool is a likert type scale consisting of 4 items: "positioning", "holding", "sucking" and "swallowing". Each item is scored between 0-2 points. The lowest and highest scores obtained from the scale are 0 and 8, respectively. Low scores indicate that breastfeeding is ineffective and high scores indicate that breastfeeding is effective.

SECONDARY OUTCOMES:
Premature infants weight (kg) | changes from birth, on the first breastfeeding day and on the breastfeeding day one week after the first breastfeeding
  The body weight will be measured every day during the oral colostrum application. on the first breastfeeding day and on the breastfeeding day one week after the first breastfeeding Weight will measure using calibrated and ten grams sensitive weighing. The measurement value will be recorded on the "preterm follow-up form" which was created by the researchers.The measurement value will be recorded on the "preterm follow-up form" which was created by the researchers.
Premature infants length/height (cm) | changes from birth, on the first breastfeeding day and on the breastfeeding day one week after the first breastfeeding
  Child length/height will obtain at every day during the oral colostrum application, on the first breastfeeding day and on the breastfeeding day one week after the first breastfeeding. Stretching tape was used for height measurement. The measurement value will be recorded on the "preterm follow-up form" which was created by the researchers.The measurement value will be recorded on the "preterm follow-up form" which was created by the researchers.
Premature infants head circumference | changes from birth, on the first breastfeeding day and on the breastfeeding day one week after the first breastfeeding
  Premature infants head circumference will obtain at every day during the oral colostrum application, on the first breastfeeding day and on the breastfeeding day one week after the first breastfeeding. Head circumference will measure with a tape measure extending from the middle of the forehead to the farthest part in the rear of the head (premature's head around its largest area). The measurement value will be recorded on the "preterm follow-up form" which was created by the researchers.
Premature infants respiratory rate | changes from birth, on the first breastfeeding day and on the breastfeeding day one week after the first breastfeeding
  Premature infants respiratory rate will obtain at every day before and after the oral colostrum administration, on the first breastfeeding day and on the breastfeeding day one week after the first breastfeeding. Respiratory rate will be assesed from monitör.The measurement value will be recorded on the "preterm follow-up form" which was created by the researchers.
Premature infants heart rate | changes from birth, on the first breastfeeding day and on the breastfeeding day one week after the first breastfeeding
  Premature infants heart rate will obtain at every day before and after the oral colostrum administration, on the first breastfeeding day and on the breastfeeding day one week after the first breastfeeding. Respiratory rate will be assesed from monitör.The measurement value will be recorded on the "preterm follow-up form" which was created by the researchers.
Premature infants body temperature | changes from birth, on the first breastfeeding day and on the breastfeeding day one week after the first breastfeeding
  Premature infants body temperature will obtain at every day before and after the oral colostrum administration, on the first breastfeeding day and on the breastfeeding day one week after the first breastfeeding. Body temperature will evaluate by a thermometer placed under axillary of new-borns. The thermometer should be placed snugly in the axillary. The measurement value will be recorded on the "preterm follow-up form" which was created by the researchers.
Premature infants oxygen saturations | changes from birth, on the first breastfeeding day and on the breastfeeding day one week after the first breastfeeding
  Premature infants heart rate will obtain at every day before and after the oral colostrum administration, on the first breastfeeding day and on the breastfeeding day one week after the first breastfeeding. Respiratory rate will be assesed from monitör. The measurement value will be recorded on the "preterm follow-up form" which was created by the researchers.

CONTACTS AND LOCATIONS:
Overall Officials: Dilek Menekşe, PhD, Study Director — Sakarya University; Nursan Cinar, professor, Principal Investigator — Sakarya University; İbrahim Caner, PhD, Principal Investigator — Sakarya University; Özge Karakaya Suzan, MSc, Principal Investigator — Sakarya University Training and Research Hospital
Locations (1):
- sakarya University, Sakarya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
typically after the end of the study

REFERENCES:
- See also: Related Info — https://trialsjournal.biomedcentral.com/articles/10.1186/s13063-015-0969-6